CLINICAL TRIAL: NCT00733733
Title: A Prospective, Randomized, Open, Multicenter Study to Evaluate the Efficacy and Tolerability of Induction Therapy With a Single High-Dose Anti-T-Lymphocyte Globulin (ATG) in Renal Transplant Patients With a Kidney From a Non-Heart-Beating Donor and Tacrolimus, Mycophenolate Mofetil, and Steroids as Basic Immunosuppression.
Brief Title: Anti-T-Lymphocyte Globulin (ATG) in Renal Transplantation of Kidneys With a Non-Heart-Beating (NHB) Donor
Acronym: ATG
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Collaborators: Erasmus Medical Center (Other); Maastricht University (Other); Leiden University Medical Center (Other); UMC Utrecht (Other); University Medical Center Groningen (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Prof. Dr. A.J. Hoitsma, UMC St Radboud Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Euro-NHB
Record Dates: First submitted 2008-08-12; First posted 2008-08-13 (Estimated); Last update posted 2008-08-13 (Estimated); Status verified 2008-08

CONDITIONS: Renal Transplant Patients; Recipients of a Kidney From a Non-Heart-Beating Donor
Keywords: kidney; transplantation; non-heart-beating donor; delayed graft function; Antithymocyte globulin; ischemia-reperfusion damage
MeSH Terms: conditions — Delayed Graft Function

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ATG (Active Comparator): One gift of ATG Fresenius (9 mg/kg body weight) intravenously during the transplantation procedure. ATG is given in addition to standard immunosuppressive treatment (tacrolimus/MMF/prednisolone)
  Interventions: Drug: ATG Fresenius
- Control (No Intervention): Standard immunosuppressive treatment for renal transplantation including tacrolimus/MMF/prednisolone without ATG treatment.

INTERVENTIONS:
Drug: ATG Fresenius — One gift of ATG Fresenius (9 mg/kg body weight) intravenously during the transplantation procedure. ATG is given in addition to standard immunosuppressive treatment (tacrolimus/MMF/prednisolone)
  Arms: ATG

SUMMARY:
One of the greatest problems in renal transplantation is the shortage of donor kidneys. Kidneys of non-heart-beating donors (NHB) are a possible solution, but transplantation is accompanied with a high percentage of acute renal failure, caused by ischemia-reperfusion injury. The increased ischemia-reperfusion injury results in an increased immune activation, which can lead to more injury of the kidney and additional acute rejections. The hypothesis of this trial is that ischemia-reperfusion injury can be diminished by ATG. ATG could have additional favourable effects. To investigate this half of the patients is treated with additional ATG to the standard immunosuppressive treatment. Calcineurin inhibitors are not diminished during the first days after transplantation to investigate whether ATG has special effects on ischemia-reperfusion injury.

ELIGIBILITY:
Inclusion Criteria:

* Non-heart-beating-donors (Maastricht III/IV)
* Female patients of childbearing age agree to maintain effective birth control practice during the study.

Exclusion Criteria:

* Pregnant or lactating women at the time of randomization.
* Patients and donors are ABO incompatible.
* Women having had >3 pregnancies (including abortions if no consistent data on PRA or anti-donor antibodies are available).
* Patients with hypersensibility to rabbit proteins, previous treatment with rabbit IgG, or known intolerance to any component of basal immunosuppression.
* Patients with leukocytes <3,000/mm3 and/or platelets <50,000/mm3 before initiation of transplant.
* Patients, who are HIV positive.
* Patients subjected to previous transplants or candidates for multiple transplants (e.g. SKP).
* Patients, who are unlikely to comply with the visit schedule in the protocol and patients who cannot communicate reliably with the investigator.
* Patients with pulmonary oedema or with other signs of overhydration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2008-01; Primary Completion 2010-01 (Estimated); Study Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of initial delayed graft function (defined as need for dialysis) | Within three months after transplantation

SECONDARY OUTCOMES:
Duration of initial delayed graft failure | Within 3 months after transplantation
Incidence of primary never-functioning grafts | Within 3 months after transplantation
Incidence of acute rejections (biopsy proven) | Within 3 months after transplantation
Renal function as determined by MDRD | At 1, 2, 3 months after transplantation
Proteinuria | At 1, 2, 3 months after transplantation
Percentage of patients with arterial hypertension | At 3 months after transplantation
Percentage of patients with antihypertensive drugs (and the number of different classes of antihypertensive drugs) | At 3 months after transplantation
Percentage of hyperlipidemic patients | At 3 months after transplantation
Percentage of post transplant diabetes mellitus | During 3 months after transplantation
Incidence of cytomegalovirus infection | During 3 months after transplantation
Incidence of tumours/PTLD | At 3 months after transplantation
Patient and graft survival | At 3 months after transplantation
Incidence of other infections | During 3 months after transplantation
Microalbuminuria | At 1, 2, 3 months after transplantation

CONTACTS AND LOCATIONS:
Overall Officials: andries hoitsma, prof.dr., Principal Investigator — UMC St Radboud Hospital, Nijmegen, the Netherlands
Locations (1):
- UMC St Radboud Hospital, Nijmegen, Netherlands